CLINICAL TRIAL: NCT05959837
Title: Usability of the Adapted Rower for People With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Regan, Clinical Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00129966
Record Dates: First submitted 2023-07-10; First posted 2023-07-25 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Intervention Arm (Experimental): Exercise intervention with adaptive rower
  Interventions: Other: Adaptive Rowing Exercise

INTERVENTIONS:
Other: Adaptive Rowing Exercise — Participants will perform two bouts of rowing exercise each with a 2-minute warm up and cool down in addition to the following: (1)10 minutes of steady state rowing with goals to achieve moderate intensity exertion levels, followed by a variable rest period to return exertion and heart rate to initial levels, (2) 10 minutes of interval rowing alternating between one minute of low-moderate intensity and 30 seconds of moderate-vigorous intensity.

SUMMARY:
The goal of this clinical trial is to examine usability of a locally built adaptive rower for people with spinal cord injury using an established and tested design.

The main questions it aims to answer are:

1. What exercise intensity of activity do users achieve on the rower for steady state and interval rowing plans?
2. What assistance is required for setup and usage of the adaptive rower?
3. What do users think about the ease of use and what is their satisfaction with the adaptive rower?

Participants will complete a one-time exercise session with two adaptive rower bouts (10-15 minutes each) with a rest period in between.

DETAILED DESCRIPTION:
A single group rolling prospective cohort study with a target of 15 participants will evaluate the initial design prototype using the an existing adaptive rower design. Participants will have one visit to the University of South Carolina Rehabilitation lab. Participants will receive an orientation to the rowing machine and available handle, grip and trunk support options. Training will be provided in proper rowing technique and use of the rate of perceived exertion scale. Participants will be fitted with a heart rate monitoring device and resting heart rate established. Participants will perform two bouts of rowing exercise each with a 2-minute warm up and cool down in addition to the following: (1)10 minutes of steady state rowing with goals to achieve moderate intensity exertion levels, followed by a variable rest period to return exertion and heart rate to initial levels, (2) 10 minutes of interval rowing alternating between one minute of low-moderate intensity and 30 seconds of moderate-vigorous intensity. Participants heart rate will be monitored and recorded throughout the testing period, with rate of perceived exertion at start, midpoint and end of steady state period, and at start, at each interval, and at end in interval period.

ELIGIBILITY:
Inclusion Criteria:

* use a wheelchair for mobility,
* can perform the rowing motion with their arms
* have enough grip strength to maintain grip on the rower handle with or without grip assist straps
* are cleared to exercise through the electronic physical readiness questionnaire or physician release

Exclusion Criteria:

* current self-reported pressure wounds
* pain with rowing motion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Heart Rate, (beats per minute), mean and range at rest, mean and range during steady state portion, mean and range during interval portion | During Exercise intervention
  Heart rate will be recorded at rest and throughout the exercise intervention using a polar heart rate monitor and actigraph.
Rate of Perceived Exertion (RPE)-Borg 6-20 Scale | During Exercise intervention
  RPE will be verbally stated by participant and recorded by study personnel at beginning, mid and end of steady state portion, and at each interval for interval exercise. (RPE, 6-20, higher means higher intensity)
Pain Scale (0-10 visual analog scale, higher means worse pain ) and body location of pain verbalized by participant and recorded by study personnel | During Exercise intervention
  participant complaints of discomfort or pain verbally stated along with location
Physical Activity Enjoyment Scale (Short); average score (1-5) | Immediately after the intervention
  A 4 item Likert scale survey to evaluate the enjoyment of the activity (1-5, higher means better outcome)
System Useability Scale, average score (1-5) | Immediately after the intervention
  A ten question Likert scale survey to evaluate a system for ease of use (1-5, higher means better outcome)
Pain Scale (0-10 visual analog scale, higher means worse pain ) and body location of pain | Two days post intervention
  participant complaints of discomfort or pain with free form location on web survey

SECONDARY OUTCOMES:
Exercise Time (minutes and seconds): recorded by study personnel | during exercise intervention
  Steady State Portion: Total Exercise Time; Interval Portion: Exercise time for each interval
Rest Time minutes and seconds: recorded by study personnel | during exercise intervention
  Steady State Portion: duration for each rest break; Interval Portion: duration for each rest break
Type of Rower Handle Used | Immediately after the intervention
  standard row, bicycle, free handles, recorded by study personnel
Grip Assist Used | Immediately after the intervention
  none, hook, velcro, combined; recorded by study personnel
Trunk Assist Used | Immediately after the intervention
  none, corset support, backpack harness; recorded by study personnel
Assistance Provided at Setup | Immediately after the intervention
  minimum, moderate, maximum with description; recorded by study personnel

OTHER OUTCOMES:
Recommendations for changes | Immediately after the intervention
  Free form comments from participants on any changes to rower design, setup or exercise protocols

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin Ginis KA, van der Scheer JW, Latimer-Cheung AE, Barrow A, Bourne C, Carruthers P, Bernardi M, Ditor DS, Gaudet S, de Groot S, Hayes KC, Hicks AL, Leicht CA, Lexell J, Macaluso S, Manns PJ, McBride CB, Noonan VK, Pomerleau P, Rimmer JH, Shaw RB, Smith B, Smith KM, Steeves JD, Tussler D, West CR, Wolfe DL, Goosey-Tolfrey VL. Evidence-based scientific exercise guidelines for adults with spinal cord injury: an update and a new guideline. Spinal Cord. 2018 Apr;56(4):308-321. doi: 10.1038/s41393-017-0017-3. Epub 2017 Oct 25. PMID 29070812
- [Background] Farkas GJ, Gorgey AS, Dolbow DR, Berg AS, Gater DR Jr. Energy Expenditure, Cardiorespiratory Fitness, and Body Composition Following Arm Cycling or Functional Electrical Stimulation Exercises in Spinal Cord Injury: A 16-Week Randomized Controlled Trial. Top Spinal Cord Inj Rehabil. 2021;27(1):121-134. doi: 10.46292/sci20-00065. PMID 33814890
- [Background] Sawatzky B, Herrington B, Choi K, Ben Mortenson W, Borisoff J, Sparrey C, Laskin JJ. Acute physiological comparison of sub-maximal exercise on a novel adapted rowing machine and arm crank ergometry in people with a spinal cord injury. Spinal Cord. 2022 Aug;60(8):694-700. doi: 10.1038/s41393-022-00757-2. Epub 2022 Feb 3. PMID 35110695
- [Background] Wong RN, Stewart AL, Sawatzky B, Laskin JJ, Borisoff J, Mattie J, Sparrey CJ, Mortenson WB. Exploring exercise participation and the usability of the adaptive rower and arm crank ergometer through wheelchair users' perspectives. Disabil Rehabil. 2022 Jul;44(15):3915-3924. doi: 10.1080/09638288.2021.1894245. Epub 2021 Mar 17. PMID 33730952
- [Background] Hansen RK, de Wit JLJ, Samani A, Laessoe U, Figlewski K, Larsen RG. Wheelchair-modified ergometer rowing exercise in individuals with spinal cord injury: a feasibility, acceptability, and preliminary efficacy study. Spinal Cord Ser Cases. 2022 Apr 30;8(1):48. doi: 10.1038/s41394-022-00518-6. PMID 35487894